CLINICAL TRIAL: NCT00545870
Title: A Randomized, Double-masked Study With Intraocular Bevacizumab Compared With Intravitreal Ranibizumab in Patients With Persistent Diabetic Macular Edema or Persistent Active Neovascularisation Following Lasercoagulation
Brief Title: Bevacizumab Versus Ranibizumab for Diabetic Retinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ursula Schmidt-Erfurth, M.D. (Other)
Responsible Party: Sponsor-Investigator, Ursula Schmidt-Erfurth, M.D., Head of Department, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 238/2006
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Bevacizumab treatment
  Interventions: Drug: bevacizumab
- B (Active Comparator): Ranibizumab treatment
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: bevacizumab — intravitreal application
  Arms: A
Drug: Ranibizumab — intravitreal application
  Arms: B

SUMMARY:
Treatment of diabetic macular edema with perifoveal focal/grid laser coagulation was found to be effective saving the visual acuity only in 50% of patients and only 3-14% of treated patients had an improved visual acuity postoperatively. The decent results of lasercoagulation are associated with potential side effects, as focal scotomas, change of color discrimination and development of epiretinal gliosis. The frequency of perifoveal laser treatments is anatomically limited in case of diabetic macular edema: after application of about 350 coagulates there is no possibility to repeat the laser treatment perifoveolar without creating confluent lasercoagulates and causing significant scotomas. In case of persistence of edema in spite of complete perifoveal grid coagulation, no standard therapy exists. Some previous studies investigated the effect of steroids in patients with diabetic macular edema unresponsive to grid laser photocoagulation, but the benefit on the visual acuity was only temporary and the intravitreal application was associated with significant side effects as cataract progression (up to 50%) and ocular hypertension (up to 20%).

In the Diabetic Retinopathy Study the 4-years rate for severe vision loss in patients with high-risk retinopathy was 20.4 %. In cases of proliferative retinopathy, panretinal (scatter) photocoagulation can reduce the risk for development of high-risk retinopathy by 50% over 6 years. When panretinal lasercoagulation is initiated, about 2000 laser spots are equally distributed in all four quadrants. Since panretinal photocoagulation bares risks like loss of field of vision, central vision reduction and loss of colour vision, this treatment can not be continued unlimited.

In cases of persisting neovascularisations in spite of panretinal photocoagulation, no evidence based therapy exists. There is a high risk for intravitreal bleeding, rubeosis, secondary glaucoma with severe vision loss. When fibrovascular proliferation leads to retinal detachment, vitreo-retinal surgery might be indicated.

Now we know that vascular endothelial growth factor (VEGF) is the major angiogenic stimulus responsible for increase of vasopermeability, cellproliferation and angiogenesis in diabetic retinopathy (DRP). Several studies, evaluating VEGF levels in vitreous, have indicated a role for VEGF in diabetic macular edema: vitreous samples of patients with diabetic macular edema contain elevated VEGF concentration and VEGF injected in experimental studies results in breakdown of the blood-retina barrier.

There is increasing evidence for a therapeutic role of anti-VEGF drugs not only in age-related macular degeneration but also in other diseases as in diabetic macular edema. Intravitreal injections have become the most favored treatment procedure for administering anti-VEGF drugs.

The side effects and the decent results of laser treatment on the visual acuity in diabetic macular edema led to studies using anti-VEGF therapy. Unpublished study results on the aptamer pegaptanib (Macugen™) are promising. A study using the antibody fragment Ranibizumab (Lucentis™) in patiens with diabetic macula edema is in progress. Ranibizumab is now approved to be used as an intravitreal injection.

Currently there is one additional anti-VEGF drug already on the market: Bevacizumab (Avastin™), which has approved as intravenous infusion for the treatment of metastatic colo-rectal cancer. Previous studies have shown that systemic use of Bevacizumab (Avastin™) can obtain very promising results on patients with choroidal neovascularisation (CNV) by age-related macular degenetration. This drug, a monoclonal full-length antibody, designed to bind all isoforms of VEGF is a large molecule. But case reports in patients with CNV caused by age-related macular degeneration and with macular edema from central retinal vein occlusion indicate that intravitreally given Bevacizumab (Avastin™) is effective in diseases originating from the choroids and the retina, too. These findings imply a sufficient penetration of the retina by Bevacizumab (Avastin™).

Based on these new findings and the important role of VEGF in diabetic retinopathy, we propose a pilot study for treatment of persistent diabetic macular edema or persisting active neovascularistaions following lasercoagulation with intravitreally administered Bevacizumab (Avastin™) or Ranibizumab (Lucentis™).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with type 1 or type 2 diabetes mellitus
* HbA1C between 6% and 9 %.
* Patients with persistent diabetic macular edema with center involvement following completed grid lasercoagulation in the study eye
* Patients with persistent active neovascularisations following completed panretinal lasercoagulation (at least 2000 spots) in the study eye
* Last perifoveolar laser treatment 3 months before study entry
* Central macular thickness (macular edema) of at least 300 - 550 microns in the central subfield as measured by OCT
* Not eligible for any currently approved treatments or experimental protocols
* Best corrected visual acuity, using ETDRS charts, of 20/25 to 20/200 (Snellen equivalent) in the study eye
* Patients with decrease in vision in the study eye due to foveal thickening from diabetic macular edema and not to other causes, in the opinion of the investigator

Exclusion Criteria:

* A condition that would preclude a patient for participation in the study in opinion of investigator, e.g., unstable medical status including glycemic control and blood pressure
* History of systemic corticosteroids within 3 months prior to randomization or topical, rectal or inhaled corticosteroids in current use more than 3 times per week
* Panretinal laser photocoagulation within the past 3 months or macular laser photocoagulation within the past 3 months in the study eye
* Previous treatment with intravitreal or sub-Tenon triamcinolone within the past 3 months in the study eye
* Previous participation in clinical trial involving anti-angiogenic drugs (pegabtanib sodium, ranibizumab, anecortave acetate, protein kinase C inhibitor, etc.)
* History of submacular surgery or other surgical intervention for diabetic macular edema except grid lasercoagulation in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To investigate the change in macular edema and the absolute change in visual acuity. To investigate the change of neovascularisation. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, MD, Principal Investigator — Dep. of Ophthalmology, Medical University of Vienna
Locations (1):
- Department of Ophthalmology, Medical University of Vienna, Vienna, Vienna, Austria